CLINICAL TRIAL: NCT05027503
Title: Investigation of the Effectiveness of the Hippotherapy Simulator Added to Respiratory Physiotherapy in Children and Adolescents with Cystic Fibrosis
Brief Title: Effectiveness of the Hippotherapy Simulator in Children and Adolescents with Cystic Fibrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Betül Çınar, Lecturer, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IUCbcinar01
Record Dates: First submitted 2021-08-19; First posted 2021-08-30 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2024-05

CONDITIONS: Cystic Fibrosis in Children
Keywords: cystic fibrosis; hippotherapy simulator; pulmonary functions; sputum expectoration; functional capacity; 6-Minute Walk Test; Postural stability; motor performance; respiratory physiotherapy
MeSH Terms: conditions — Cystic Fibrosis | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group (Active Comparator): Home-based respiratory physiotherapy will be applied twice a day and every day of the week for 8 weeks
  Interventions: Other: Respiratory Physiotherapy
- Training Group (Experimental): In addition to home-based respiratory physiotherapy, 30 min exercises with the hippotherapy simulator will be done.
  Interventions: Other: Exercise with hippotherapy simulator; Other: Respiratory Physiotherapy

INTERVENTIONS:
Other: Exercise with hippotherapy simulator — 30-minute (5 min warm-up+20 min exercise+5 min cool-down) center-based exercise with the hippotherapy simulator will be done 2 days a week for 8 weeks.
  Arms: Training Group
Other: Respiratory Physiotherapy — Respiratory physiotherapy includes breathing control (5x2), diaphragmatic breathing exercises (5x2), thoracic expansion exercises (5x2), incentive spirometer (5x2), opep device (5x2), postural drainage and percussion and cough improvement techniques (10 min). Home-based respiratory physiotherapy will be applied twice a day and every day of the week for 8 weeks.

SUMMARY:
Cystic fibrosis (CF) is a genetic disease that affects many organs and systems, especially respiratory system problems due to lung damage. Patients often have difficulty in removing the sticky and viscous secretion that accumulates in the respiratory tract, and the risk of mortality increases with the development of respiratory failure. In patients with CF, exercise capacity, peripheral muscle strength, core endurance, flexibility, postural stability, physical activity level, and quality of life also decrease secondarily. Recently published guidelines recommend respiratory physiotherapy for coping with CF-related symptoms and recommend referral of patients to physical activity and exercise.

Hippotherapy simulator is a mechanical exercise tool that imitates the walking movement of a real horse and is used to increase physical fitness parameters.

This study aims to show the effects of exercises performed with a hippotherapy simulator in addition to respiratory physiotherapy on physical fitness, sputum production, physical activity and quality of life of children with CF.

ELIGIBILITY:
Inclusion Criteria:

* Be in the 8-14 age range
* To be diagnosed with cystic fibrosis according to the American Cystic Fibrosis Association consensus report criteria
* Having mild (FEV1 ≥ 70% predictive) lung disease according to the disease severity classification in the annual report of the American Cystic Fibrosis Society
* To be able to produce phlegm

Exclusion Criteria:

* Contracture or deformity,
* History of diagnosed orthopedic problems affecting mobility or musculoskeletal surgery
* History of previous lung or liver transplant
* Have diagnosed vision, hearing, vestibular or neurological problems that may affect balance,
* History of hospitalization in the last 1 month
* Patients who have participated in any exercise training program in the last 6 months

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2021-12-19 (Actual); Primary Completion 2024-02-19 (Actual); Study Completion 2024-05-26 (Actual)

PRIMARY OUTCOMES:
Forced Vital Capacity (FVC) | 8 weeks
  Pulmonary Function Test
Forced Expiratory Volume in 1 second (FEV1) | 8 weeks
  Pulmonary Function Test
Tiffeneau ratio (FEV1/FVC) | 8 weeks
  Pulmonary Function Test
Peak Expiratory Flow (PEF) | 8 weeks
  Pulmonary Function Test
Distance covered in six minute walk test | 8 weeks
  Functional Capacity
Postural stability test score in Biodex Balance System SD | 8 weeks
  Postural Stability
Limits of stability test score in Biodex Balance System SD | 8 weeks
  Postural Stability

SECONDARY OUTCOMES:
Biering Sorenson Test | 8 weeks
  Core Muscles Endurance
Lateral Bridge Test | 8 weeks
  Core Muscles Endurance
Trunk Flexion Test | 8 weeks
  Core Muscles Endurance
m. quadriceps strength | 8 weeks
  Peripheral Muscle Strength
Amount of sputum expelled (gr) | 8 weeks
  Sputum amount
Ease of expectoration | 8 weeks
  Subjective assessment that evaluates "how hard the person has during sputum production" with a visual analog scale (0-10 point). A high score means that it is easy to sputum.
Sense of chest congestion | 8 weeks
  Subjective evaluation method questioning "sense of chest congestion" with visual analog scale (0-10 point). A higher score indicates greater sense of chest congestion.
Sit and reach test | 8 weeks
  Flexibility
Physical Activity Questionnaire for Children (PAQ-C) | 8 weeks
  Physical Activity Level. As a result of the 9-item questionnaire, 1 means lowest and 5 means highest physical activity level.
Cystic Fibrosis Questionnaire Revised (CFQ-R) | 8 weeks
  Quality of Life Assessment. In this questionnaire, which consists of 35 questions, the total score is 100, and a higher score indicates a better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Betül Çınar, Principal Investigator — Istanbul University - Cerrahpasa
Locations (1):
- Bezmialem Vakif University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No